CLINICAL TRIAL: NCT00726947
Title: Aging Venous Thrombi With Ultrasound Elasticity Imaging
Brief Title: Ultrasound Elasticity Imaging of Venous Thrombi
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Rubin, M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 0040239; NIH ROI HL 78656-01A1
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ultrasound imaging of Acute DVT (deep vein thrombosis)
  Interventions: Procedure: Ultrasound
- 2 (Experimental): Ultrasound imaging of Chronic DVT (deep vein thrombosis)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound imaging of Acute DVT
  Arms: 1
Procedure: Ultrasound — Ultrasound imaging of Chronic DVT
  Arms: 2

SUMMARY:
The purpose of this study is to see if the investigators can use ultrasound imaging to determine the type of clots in patients to help better manage their care.

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) is a blood clot and is a common illness that can result in pain and death if not recognized and treated well. Death can occur when the venous clots break off and form pulmonary emboli (PE), which can block the arteries of the lungs. DVT and PE most often complicate the course of sick patients but may also affect healthy persons. DVT can also be a chronic disease. In those instances in which DVT and PE develop, in addition to the death risk, hospitalization is drawn out and healthcare costs are increased. Therefore, the purpose of this study is to see if we can use ultrasound imaging to determine the type of clots in patients to help better manage their care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who have a diagnosis of chronic DVT that is at least 2 weeks old and are free from an acute DVT on top of your chronic DVT.
* Male and female patients who have been diagnosed with an acute blood clot by the Diagnostic Vascular Lab and w/symptoms occurring within the previous 2 weeks.
* Patients under the age of 18 who give assent (permission) and whose parents give consent.
* Adult patients who give consent.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2002-12; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine if ultrasound imaging will aid in the diagnosis and classification of venous blood clots | approximately one year

SECONDARY OUTCOMES:
Follow-up with subjects who have been diagnosed with Acute DVT to see if they develop post-thrombotic syndrome (PTS) | first year following diagnosis of acute DVT

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No